CLINICAL TRIAL: NCT06390462
Title: Adolescent Depression Treatment Pathways in Primary Care - a Longitudinal Cohort Study Describing Naturalistic Flow of Treatment and Evaluating Effectiveness and Cost-effectiveness of Interpersonal Counseling Compared to Treatment as Usual
Brief Title: Adolescent Interpersonal Counseling in Primary Care
Status: Recruiting | Type: Observational
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Strategic Research Council of Finland (Unknown); University of Helsinki (Other); University of Eastern Finland (Other); Tampere University (Other)
Responsible Party: Sponsor
Other Study IDs: 1271/6.02.03/2024
Record Dates: First submitted 2024-03-19; First posted 2024-04-30 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Depressive Symptoms Mild to Moderate in Severity; Major Depressive Disorder
Keywords: adolescent; depression; prospective; cohort study; interpersonal counseling; prevention; therapy; effectiveness; cost-effectiveness; predictor; economic evaluation
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Therapeutics; Methods

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents with sustained depression: PHQ-9-A ≥ 10 at least twice in a 6 months follow-up
  Interventions: Behavioral: Interpersonal counseling; Behavioral: Treatment as usual; Other: No support, intervention or other treatment

INTERVENTIONS:
Behavioral: Interpersonal counseling — A structured psychotherapeutic intervention to prevent depression or treat mild to moderate depression. IPC-A is a brief, individual-based intervention (3-8 sessions). The focus is on interpersonal relations as a factor of resilience in depressive symptoms. IPC-A is a shorter form of IPT-A, developed by prof. Myrna Weissman and team.
Behavioral: Treatment as usual — Any other behavioral or medical support or depression indicated by depressive symptoms or depression. This is based on adolescent, caretaker and professional's report.
Other: No support, intervention or other treatment — The group will comprise those adolescents who report sustained depression but do not seek or receive support over 6 months of follow-up based on adolescent and caretaker's report

SUMMARY:
The demand for prevention and treatment of adolescent depression has rapidly increased over years. A national project to improve treatment of adolescent depression in primary care has taken place in Finland starting 2020.

The goal of this prospective observational cohort study is to describe pathways to mental health services in adolescents with depressive symptoms. The main questions it aims to answer are:

* Do young people reporting depressive symptoms have equal access to treatment?
* How is it best to recognize those adolescents who will benefit from IPC-A?

Adolescents who participate in the study will

* complete a survey on protective and risk factors of depression three times over 6 months
* report possible depressive symptoms every two weeks over 6 months
* report whether they needed and received help, motivation for treatment, and benefits and harms from treatment

We will also collect

* information from one of caretakers with two surveys within 6 month- intervals on their view on adolescent's need for support, strengths and risks, and benefits and harms from treatment where applicable
* where applicable, from the professional who provided support after the intervention on their training and competence, as well as content of and response to treatment
* register data to estimate overall provision and cost of social welfare and health care services one year preceding the study and over 2 to 10 years after the observation period

Researchers will compare an intervention that is new in Finland, adolescent interpersonal counseling (IPC-A), to other treatments of depression, to see if it is equal to or better than other treatments of depression.

DETAILED DESCRIPTION:
Background: Implementation of evidence-based interventions is one of the proposed responses to increased demand for prevention and treatment of adolescent depression. A national implementation of adolescent interpersonal counseling (IPC-A) has taken place in Finland starting 2020. While the efficacy of interpersonal psychotherapy (IPT-A) as an intervention to treat depression of adolescents is well established, the effectiveness and cost-effectiveness of the shorter adaptation, IPC-A, remains open. Investigators present a protocol for an evaluation of pathways to mental health services of depressed adolescents and a prospective, observational community-based cohort study to estimate the effectiveness and cost-effectiveness of IPC-A, as compared to adolescents with sustained depression with treatment as usual or no treatment.

Methods: The cohort will include grade 7 to 9 adolescents (13-16-year-olds) in selected Finnish schools, excluding adolescents with preceding treatment of depression. A universal prospective evaluation of adolescents in a 6-month follow-up will provide information on the proportion of adolescents a) with sustained depression over the follow-up period (Patient Health Questionnaire 9 items, PHQ-9 ≥ 10) in two measurements over 6 months), b) with a self-reported need for support due to depressive symptoms, and c) with a therapeutic intervention. The investigators will describe the treatment received (number of sessions, therapeutic content) based on reports from adolescents, caretakers, and therapists, as well as electronic patient records. The primary outcome measure will be the proportion of adolescents who will receive specialized psychiatric services by 12 months after baseline. Secondary outcome measures comparing three groups as defined at 6 months (IPC-A, treatment as usual (TAU), or no treatment group). They will include proportion of adolescents who received any support by 12 months after baseline, and longitudinal changes in PHQ-9-A scores by 12 months. Cost-effectiveness will be evaluated using survey data at 12 months, and an economic evaluation using register data and information on service use 12 months before and 2 and 10 years after baseline. Collection of survey data is expected to start in March 2024 and is set to finish in May 2025.

Discussion: The study will describe need for, pathways to, and content of social and health services for depressed adolescents. Benefits and harms of treatment and the national implementation will be observed. The results can improve detection and equal access to care, and inform decision-makers about the best practices for prevention, including utility of the implementation of IPC-A.

ELIGIBILITY:
Inclusion Criteria:

* we will include all adolescents attending grades 7 to 9 in selected schools with on informed consent

Exclusion Criteria:

* psychiatric care within the past 12 months or receiving a psychosocial intervention (psychotherapy, IPC-A, any other therapy of support) during the 12 months before baseline,
* an inability to reliably understand the Finnish, Plain Finnish, Swedish, or English versions of the survey, or
* an adolescents' or caretakers' report of a need for exclusion, such as another medical condition - including a mental disorder - requiring acute current treatment or support.

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents attending grades 7 to 9 (13 to 16 years) in selected schools
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2039-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of adolescents referred to specialized psychiatric services | From baseline to 12 months
  Proportion of adolescents in each three groups with sustained depressive symptoms by 6 months who receive specialized psychiatric services by 12 months

SECONDARY OUTCOMES:
Proportion of adolescents who received any social welfare or health care services | Up to 10 years after baseline
  Data collected from adolescent and caretaker's surveys and registers
longitudinal changes in PHQ-9-A score | 2 weeks
  Longitudinal changes in biweekly PHQ-9-A scores over 6 months; PHQ-9-A 10 items, 0 to 3, higher score more depression

OTHER OUTCOMES:
Loneliness | No time frame
  One item: Do you feel lonely? yes/no
Experiences of Social Inclusion Scale | No time frame
  10 items, 0 to 4, higher score more inclusion
The child-friendly EuroQol-5 dimensions questionnaire | The same day
  EQ-5D-Y, 5 items 0 to 2; a VAS scale, higher score more functional
Generalized Anxiety Disorder Scale-7 | 2 weeks
  GAD-7, 7 items 0 to 3, higher score more anxiety
The Short Warwick-Edinburg Mental Wellbeing Scale | 2 weeks
  SWEMWBS, 7 items for positive mental health 0 to 4, higher score more positive mental health
Young Person's Clinical Outcomes in Routine Evaluation-Outcome Measure | 1 week
  YP-CORE; 10 items 0 to 4, higher score better outcome
3x10D life situation assessment tool | No time frame
  3x10-Dx, 10 items 0 to 0, higher score better life situation
Harmful behavior: Alcohol and substance use, self-harming behavior | Ever, past 30 days
  Questions yes/no, open field

CONTACTS AND LOCATIONS:
Overall Officials: Outi Linnaranta, MD, PhD, Principal Investigator — Finnish Institute for Health and Welfare
Locations (4):
- Finland (4):
  - The wellbeing services county of Kanta-Häme, Hämeenlinna
  - Finnish Institute for Health and Welfare, Helsinki
  - The wellbeing services county of Central Finland, Jyväskylä
  - The wellbeing services county of North Ostrobothnia, Oulu

IPD SHARING:
Plan to Share IPD: Yes
Mauri Marttunen and Klaus Ranta: effectiveness and psychometrics; Johanna Lammintakanen: cost-effectiveness and economic evaluation; Jari Lahti: motivation to treatment; Erkki Heinonen: Therapist competence and outcome
Supporting Information: Study Protocol, SAP, ICF
Time Frame: First baseline IPD available from fall 2025 for 10 years, final economic evaluation data will be stored from 2039 for 10 years
Access Criteria: Data access is restricted by user roles with permission of PI (Outi Linnaranta), and all data will be pseudonymized. Sensitive register data including person IDs will be managed using the Findata Kapseli service.
URL: https://stnimagine.fi/tyopaketti-4-vaikuttavuusseuranta/

REFERENCES:
- See also: Description in Finnish and in English about the study, participant informed consent (adolescent, caretaker, professional) — https://stnimagine.fi/tyopaketti-4-vaikuttavuusseuranta/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT06390462/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT06390462/ICF_001.pdf